CLINICAL TRIAL: NCT07124065
Title: Differentiation of Benign From Malignant Thyroid Nodules Using Diffuse Reflectance Spectroscopy
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 08/H0719/37
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Thyroid Cancer; Nodule Solitary Thyroid
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients undergoing surgery for thyroid nodules
  Interventions: Diagnostic Test: Diffuse reflectance spectroscopy

INTERVENTIONS:
Diagnostic Test: Diffuse reflectance spectroscopy — Spectral data collection with diffuse reflectance spectroscopy

SUMMARY:
Patients with thyroid nodules are currently investigated with ultrasound with or without biopsy. Despite these investigations, a subset of patients remain "indeterminate" whereby a cancer can neither be diagnosed nor ruled out - these patients will usually be recommended to undergo diagnostic surgery. This study aims to assess a new technique called diffuse reflectance spectroscopy to determine if this can differentiate between benign and cancerous nodules, particularly in these indeterminate cases.

DETAILED DESCRIPTION:
Diffuse reflectance spectroscopy is an imaging technique which is conducted via a probe that is placed into direct contact with the tissue. This probe emits light, and simultaneously measures the light reflected back - differences in this reflected light can provide valuable information which may be able to differentiate cancerous from non-cancerous tissue. Several previous studies have proven this technique useful in other tissues, such as the stomach and oesophagus - this study therefore aims to assess its utility for thyroid nodules

The spectroscopic probe is used on the tissue that has already been taken from the body as part of the operation, not on the inside of the body itself. The tissue samples being removed will routinely be sent for microscopic analysis to inform the surgeon about the type of tissues present in the area of the body being operated on. The research team will be in the operating theatre and use the optical probe on the tissue samples.The probe will only be used on the tissue after it has been removed by the surgeon; therefore, the probe will not impact on the operation.

The overall aim of the study is to determine if this probe is able to differentiate which nodules are benign and which are cancerous.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing surgery for thyroid nodules
* age 18 years and over
* radiological/cytological assessment of nodule pre-operatively

Exclusion Criteria:

* declined consent
* lack capacity
* emergency surgery
* re-operative surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery for thyroid nodules at Hammersmith Hospital, UK
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Cancer diagnosis | Single time point only (intra-operative data collection)
  To determine if DRS can differentiate cancerous nodules from benign from spectral data

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No